CLINICAL TRIAL: NCT00476541
Title: NOPHO-AML 2004 Study for Children With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOPHO-AML 2004
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Children; Gemtuzumab ozogamicin; Stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Gemtuzumab 5 mg / m2 two courses with three week interval
  Interventions: Drug: Gemtuzumab ozogamicin
- 2 (No Intervention): No further therapy

INTERVENTIONS:
Drug: Gemtuzumab ozogamicin — Two courses of Gemtuzumab vs. no further therapy
  Other Names: Mylotarg
  Arms: 1

SUMMARY:
The overall objective is to improve the cure rate of children with newly diagnosed acute myeloid leukemia (AML) who undergo risk-adapted therapy.

Stem cell transplantation (SCT) is reserved to high-risk patients defined by cytogenetics and response to chemotherapy. The efficacy and toxicity of Gemtuzumab ozogamicin (GO, Mylotarg) will be evaluated.

DETAILED DESCRIPTION:
The overall objective is to improve the cure rate of pediatric patients with newly diagnosed acute myeloid leukemia (AML). The specific aims are as follows:

1.1 Therapeutic aims

To improve the event-free survival (EFS) of AML patients who undergo risk-adapted therapy.

To improve the overall survival (OS) by reserving stem cell transplantation (SCT) to high-risk patients based on cytogenetics and response to induction therapy.

To compare the outcome of SCT using HLA-matched sibling donor (MSD) or HLA-matched unrelated donor (MUD).

To assess the efficacy and toxicity of Gemtuzumab ozogamicin (GO, Mylotarg) as post consolidation therapy.

1.2 Biologic aims

To study minimal residual disease (MRD) levels in blood and bone marrow (BM) at defined time points and to study the prognostic impact of MRD.

To test in vitro cellular drug resistance at diagnosis and relapse, and correlate these data to background factors and clinical outcome.

To secure storage of biological material from diagnosis for future biologic studies

ELIGIBILITY:
Inclusion Criteria:

* AML as defined by the diagnostic criteria,
* Age < 19 years at time of study entry,
* Written informed consent

Exclusion Criteria:

* Previous chemo- or radiotherapy,
* AML secondary to previous bone marrow failure syndrome,
* Down syndrome (DS),
* Acute promyelocytic leukemia (APL),
* Juvenile myelomonocytic leukemia (JMML),
* Myelodysplastic syndrome (MDS),
* Fanconi anemia,
* Positive pregnancy test

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2004-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Event free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Hasle, MD, Study Chair — Department of Pediatrics, Aarhus University Hospital Skejby, Aarhus, Denmark
Locations (2):
- Denmark (2):
  - Department of Pediatrics, Aarhus University Hospital Skejby, Aarhus
  - Rigshospitalet, Copenhagen

REFERENCES:
- [Background] Lie SO, Abrahamsson J, Clausen N, Forestier E, Hasle H, Hovi L, Jonmundsson G, Mellander L, Siimes MA, Yssing M, Zeller B, Gustafsson G; Nordic Society of Pediatric Hematology and Oncology (NOPHO); AML Study Group. Long-term results in children with AML: NOPHO-AML Study Group--report of three consecutive trials. Leukemia. 2005 Dec;19(12):2090-100. doi: 10.1038/sj.leu.2403962. PMID 16304571
- [Background] Lie SO, Abrahamsson J, Clausen N, Forestier E, Hasle H, Hovi L, Jonmundsson G, Mellander L, Gustafsson G. Treatment stratification based on initial in vivo response in acute myeloid leukaemia in children without Down's syndrome: results of NOPHO-AML trials. Br J Haematol. 2003 Jul;122(2):217-25. doi: 10.1046/j.1365-2141.2003.04418.x. PMID 12846889
- [Derived] Hasle H, Abrahamsson J, Forestier E, Ha SY, Heldrup J, Jahnukainen K, Jonsson OG, Lausen B, Palle J, Zeller B; Nordic Society of Paediatric Haematology and Oncology (NOPHO). Gemtuzumab ozogamicin as postconsolidation therapy does not prevent relapse in children with AML: results from NOPHO-AML 2004. Blood. 2012 Aug 2;120(5):978-84. doi: 10.1182/blood-2012-03-416701. Epub 2012 Jun 22. PMID 22730539